CLINICAL TRIAL: NCT04450849
Title: Regenerative Potential of a Collagen Membrane Associated or Not to Bovine Bone in Class II Furcation Defects - A Randomized Clinical Trial.
Brief Title: Regenerative Potential of a Collagen Membrane Associated or Not to Bovine Bone in Class II Furcation Defects.
Acronym: RPPCMABBICFD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Sergio Luis Scombatti de Souza, Departament of Oral & Maxillofacial Surgery and Periodontology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008.1.1259.58.9
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Periodontal Diseases; Bone Diseases
Keywords: periodontal diseases; Periodontitis; periodontal regeneration
MeSH Terms: conditions — Periodontal Diseases; Bone Diseases; Periodontitis | interventions — Guided Tissue Regeneration; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Intervention Model Description: In a parallel design, 22 patients with mandibular class II furcation defects were recruited. Each defect was randomly assigned to the control group (CG - Bio-Gide® Perio, n=11) or test group (TG - Bio-Oss® Collagen + Bio-Gide® Perio, n=11). Tomographic and clinical evaluations were conducted at baseline and 12 months post-surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- collagen membrane associated to anorganic bone (Experimental): Complete debridement of the osseous defects and thorough scaling and root planing using mini curettes and ultrasonic scalers were performed. The sites were randomly selected for treatment with resorbable collagen membrane (Bio-Gide® Perio) associated to anorganic bovine bone matrix + collagen (Bio-Oss® Collagen) . The membranes were trimmed to cover the lesions and extended to the adjacent bone between 2 to 3 mm apically and laterally. They were then placed in position, 2 mm below the CEJ, and fixed in position using sling 5-0 vicryl sutures. The flaps were coronally positioned until completely covering the membranes without tension and sutured with 5-0 nylon sutures
  Interventions: Procedure: guided tissue regeneration with using an absorbable collagen membrane associated with inorganic bovine bone associated.
- collagen membrane alone (Active Comparator): Complete debridement of the osseous defects and thorough scaling and root planing using mini curettes and ultrasonic scalers were performed. The sites were randomly selected for treatment with resorbable collagen membrane (Bio-Gide® Perio). The membranes were trimmed to cover the lesions and extended to the adjacent bone between 2 to 3 mm apically and laterally. They were then placed in position, 2 mm below the CEJ, and fixed in position using sling 5-0 vicryl sutures. The flaps were coronally positioned until completely covering the membranes without tension and sutured with 5-0 nylon sutures
  Interventions: Procedure: guided tissue regeneration with using an absorbable collagen membrane associated or not with inorganic bovine bone associated with collagen matrix.

INTERVENTIONS:
Procedure: guided tissue regeneration with using an absorbable collagen membrane associated with inorganic bovine bone associated. — Dental surgical procedures that use barrier membranes to direct the growth of new bone and gingival tissue at sites with insufficient volumes or dimensions of bone or gingiva for proper function, esthetics or prosthetic restoration. Using an absorbable collagen membrane (Bio-Gide® Perio) associated with inorganic bovine bone associated with collagen matrix (Bio-Oss® Collagen).
  Other Names: GTR
  Arms: collagen membrane associated to anorganic bone
Procedure: guided tissue regeneration with using an absorbable collagen membrane associated or not with inorganic bovine bone associated with collagen matrix. — dental surgical procedures that use barrier membranes to direct the growth of new bone and gingival tissue at sites with insufficient volumes or dimensions of bone or gingiva for proper function, esthetics or prosthetic restoration. Using an absorbable collagen membrane (Bio-Gide® Perio) alone.
  Other Names: GTR
  Arms: collagen membrane alone

SUMMARY:
Periodontal disease is an infectious-inflammatory disease that accommodates the supporting and supporting tissues of the teeth, with the formation of periodontal pockets, and this destruction can generate anatomical defects in the region of bifurcation. Treatment of these lesions is a challenge for the clinician, as this area has limited access to bacterial biofilm and calculus. The surgical regenerative therapy using bone grafts and membrane may be a viable option in cases of class II furcation defects. In this context, the objective of this case series is to evaluate tomographically and clinically the treatment of class II furcation defects using an absorbable collagen membrane (Bio-Gide® Perio) associated or not with inorganic bovine bone associated with collagen matrix (Bio-Oss® Collagen).

DETAILED DESCRIPTION:
Periodontal disease is an infectious-inflammatory disease that accommodates the supporting and supporting tissues of the teeth, with the formation of periodontal pockets, and this destruction can generate anatomical defects in the region of bifurcation. Treatment of these lesions is a challenge for the clinician, as this area has limited access to bacterial biofilm and calculus. The surgical regenerative therapy using bone grafts and membrane may be a viable option in cases of class II furcation defects. In this context, the objective of this case series is to evaluate tomographically and clinically the treatment of class II furcation defects using an absorbable collagen membrane (Bio-Gide® Perio) associated or not with inorganic bovine bone associated with collagen matrix (Bio-Oss® Collagen). In a parallel design, 22 patients with mandibular class II furcation defects were recruited. Each defect was randomly assigned to the control group (CG - Bio-Gide® Perio, n=11) or test group (TG - Bio-Oss® Collagen + Bio-Gide® Perio, n=11). Tomographic and clinical evaluations were conducted at baseline and 12 months post-surgery. Clinical measurements of clinical attachment level (CAL) and probing depth (PD). Tomographical measurements of horizontal defect dimension (HDD) and vertical defect dimension (VDD) were recorded. In sequence, guided tissue regeneration surgeries were conducted: Then, bone defect were debrided, , the collagen membranes (BioGide Perio®) were trimmed to cover the osseous defects and extended 3 mm apically and laterally to the adjacent bone and sutured with absorbable suture. In the Test Group, the defects were completely filled with bovine bone + porcine collagen (BioOss Collagen®). The flaps were then coronally positioned until completely covering the membranes and sutured. Shapiro-Wilk test was used to evaluate normality of the data, and showed a normal distribution. Then, t-Test was selected for inter-group and intragroup comparisons. Trans-surgical measurements were evaluated at Baseline. The other clinical and tomographic parameters were evaluated at Baseline and 12 months. For all analyzes, p <0.05 was considered.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a diagnosis of periodontitis, Stage III and Grade A (according to the 2018 international classification criteria);
* presence of one mandibular molar with class II buccal furcation defect;
* non-smokers;
* plaque index <20%.

Exclusion Criteria:

* patients that presented systemic diseases;
* patients that had taken antibiotics in the past 6 months prior to surgical procedures;
* pregnant women or lactating mothers;
* furcation involvement in molars with periapical disease;
* cervical restorations or prosthesis closer than 1 mm to fornix.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
to evaluate clinical attachment level | The clinical periodontal parameter will be recorded at baseline (pre-intervention) and +360 days after the surgical periodontal therapy.]
  Change from Baseline in clinical attachment level at +360 days

SECONDARY OUTCOMES:
Tomographic bone gain | The Tomographic bone gain parameter will be recorded at baseline (pre-intervention) and +360 days after the surgical periodontal therapy.]
  Change from Baseline in bone gain at +360 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided